CLINICAL TRIAL: NCT06762561
Title: Prophylactic Mesh Reinforcement After Open Aortic Aneurysm Repair: a Retrospective Study
Brief Title: Prophylactic Mesh Reinforcement After Open Aortic Aneurysm Repair
Status: Recruiting | Type: Observational
Sponsor: Hôpital Fribourgeois (Other)
Responsible Party: Sponsor
Other Study IDs: 2348
Record Dates: First submitted 2024-12-31; First posted 2025-01-07 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Incisional Hernia; Aortic Aneurysm
MeSH Terms: conditions — Incisional Hernia; Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prophylactic mesh reinforcement after open aortic aneurysm repair: Patients who underwent open abdominal aortic aneurysm (AAA) repair with prophylactic retromuscular mesh reinforcement at the Fribourg Cantonal Hospital between 2019 and 2024.
  Interventions: Procedure: Prophylactic retromuscular mesh reinforcement

INTERVENTIONS:
Procedure: Prophylactic retromuscular mesh reinforcement — Prophylactic retromuscular mesh placement involves reinforcing the abdominal wall during closure after open abdominal aortic aneurysm (AAA) repair to prevent incisional hernias. This technique creates a retro-muscular space by carefully dissecting the rectus abdominis muscles from the posterior rectus sheath. A self-gripping polyester mesh or composite mesh is placed in this space, extending 4 cm beyond the midline on each side, ensuring tension-free coverage. The mesh is secured at key points, and the rectus sheaths are closed with continuous sutures. This approach leverages the anatomical integrity of the abdominal wall to reduce hernia risk without increasing postoperative complications.

SUMMARY:
The goal of this retrospective observational study is to evaluate whether prophylactic mesh reinforcement during abdominal wall closure can prevent incisional hernias (IH) in patients undergoing open abdominal aortic aneurysm (AAA) repair. The main questions it aims to answer are:

* Does mesh reinforcement reduce the incidence of incisional hernias?
* What is the frequency of associated postoperative complications? Researchers will compare the outcomes of patients who underwent mesh-reinforced closures to literature-reported outcomes for non-mesh cases to assess differences in IH incidence and complications.

Participants will:

* Undergo clinical follow-ups and abdominal ultrasounds to detect IH.
* Complete quality-of-life questionnaires (EQ-5D and PROMIS).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old) who underwent open abdominal aortic aneurysm (AAA) repair with prophylactic retromuscular mesh reinforcement between January 2019 and January 2024
* Availability of complete medical records, including preoperative history, surgical details, and postoperative follow-up data
* Attendance at a clinical follow-up examination at least one year after the procedure
* General informed consent signed for the use of medical data for research purposes

Exclusion Criteria:

* Patients with incomplete or missing medical records, including preoperative, intraoperative, or follow-up data
* Patients who required a re-laparotomy involving incision or suture of the prophylactic mesh and subsequently developed an incisional hernia.
* Patients who did not attend the required clinical follow-up examination at least one year postoperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients who underwent open abdominal aortic aneurysm (AAA) repair with prophylactic retromuscular mesh reinforcement at the Fribourg Cantonal Hospital between 2019 and 2024.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Rate of incisional hernias | january-april 2025
  Incisional hernia will be evaluated trough clinical examination and ultrasound assessement

SECONDARY OUTCOMES:
Rate of fascial dehiscence | january-april 2025
  Fascial dehiscence will be searched in the patient's records
Rate of seromas | january-april 2025
  will be searched in the patient's records
Rate of surgical site infection | january-april 2025
  will be searched in the patient's records
Rate of hematomas | january-april 2025
  will be searched in the patient's records
Operative time | january-april 2025
  will be searched in the operation protocols

CONTACTS AND LOCATIONS:
Locations (1):
- HFR Hopitaux Fribourgeois, Villars-sur-Glâne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Endo T, Miyahara K, Shirasu T, Mochizuki Y, Taniguchi R, Takayama T, Hoshina K. Risk Factors for Incisional Hernia After Open Abdominal Aortic Aneurysm Repair. In Vivo. 2023 Nov-Dec;37(6):2803-2807. doi: 10.21873/invivo.13393. PMID 37905664
- [Background] Antoniou GA, Muysoms FE, Deerenberg EB. Updated Guideline on Abdominal Wall Closure from the European and American Hernia Societies: Transferring Recommendations to Clinical Practice for Vascular Surgeons. Eur J Vasc Endovasc Surg. 2023 Jun;65(6):774-777. doi: 10.1016/j.ejvs.2023.02.009. Epub 2023 Feb 16. No abstract available. PMID 36804613
- [Background] Antoniou GA, Georgiadis GS, Antoniou SA, Granderath FA, Giannoukas AD, Lazarides MK. Abdominal aortic aneurysm and abdominal wall hernia as manifestations of a connective tissue disorder. J Vasc Surg. 2011 Oct;54(4):1175-81. doi: 10.1016/j.jvs.2011.02.065. Epub 2011 Aug 6. PMID 21820838
- [Background] DeAngelo N, Perez AJ. Hernia Prevention: The Role of Technique and Prophylactic Mesh to Prevent Incisional Hernias. Surg Clin North Am. 2023 Oct;103(5):847-857. doi: 10.1016/j.suc.2023.04.021. Epub 2023 Jun 9. PMID 37709391
- [Background] Franchi M, Ghezzi F, Buttarelli M, Tateo S, Balestreri D, Bolis P. Incisional hernia in gynecologic oncology patients: a 10-year study. Obstet Gynecol. 2001 May;97(5 Pt 1):696-700. doi: 10.1016/s0029-7844(01)01192-9. PMID 11339918
- [Background] Sorensen LT, Hemmingsen UB, Kirkeby LT, Kallehave F, Jorgensen LN. Smoking is a risk factor for incisional hernia. Arch Surg. 2005 Feb;140(2):119-23. doi: 10.1001/archsurg.140.2.119. PMID 15723991
- [Background] Goodenough CJ, Ko TC, Kao LS, Nguyen MT, Holihan JL, Alawadi Z, Nguyen DH, Flores JR, Arita NT, Roth JS, Liang MK. Development and validation of a risk stratification score for ventral incisional hernia after abdominal surgery: hernia expectation rates in intra-abdominal surgery (the HERNIA Project). J Am Coll Surg. 2015 Apr;220(4):405-13. doi: 10.1016/j.jamcollsurg.2014.12.027. Epub 2015 Jan 2. PMID 25690673
- [Background] Montalti R, Mimmo A, Rompianesi G, Serra V, Cautero N, Ballarin R, De Ruvo N, Cunningham Gerring R, Enrico Gerunda G, Di Benedetto F. Early use of mammalian target of rapamycin inhibitors is an independent risk factor for incisional hernia development after liver transplantation. Liver Transpl. 2012 Feb;18(2):188-94. doi: 10.1002/lt.22445. PMID 21987434
- [Background] Deerenberg EB, Henriksen NA, Antoniou GA, Antoniou SA, Bramer WM, Fischer JP, Fortelny RH, Gok H, Harris HW, Hope W, Horne CM, Jensen TK, Kockerling F, Kretschmer A, Lopez-Cano M, Malcher F, Shao JM, Slieker JC, de Smet GHJ, Stabilini C, Torkington J, Muysoms FE. Updated guideline for closure of abdominal wall incisions from the European and American Hernia Societies. Br J Surg. 2022 Nov 22;109(12):1239-1250. doi: 10.1093/bjs/znac302. PMID 36026550
- [Background] Wanhainen A, Van Herzeele I, Bastos Goncalves F, Bellmunt Montoya S, Berard X, Boyle JR, D'Oria M, Prendes CF, Karkos CD, Kazimierczak A, Koelemay MJW, Kolbel T, Mani K, Melissano G, Powell JT, Trimarchi S, Tsilimparis N; ESVS Guidelines Committee; Antoniou GA, Bjorck M, Coscas R, Dias NV, Kolh P, Lepidi S, Mees BME, Resch TA, Ricco JB, Tulamo R, Twine CP; Document Reviewers; Branzan D, Cheng SWK, Dalman RL, Dick F, Golledge J, Haulon S, van Herwaarden JA, Ilic NS, Jawien A, Mastracci TM, Oderich GS, Verzini F, Yeung KK. Editor's Choice -- European Society for Vascular Surgery (ESVS) 2024 Clinical Practice Guidelines on the Management of Abdominal Aorto-Iliac Artery Aneurysms. Eur J Vasc Endovasc Surg. 2024 Feb;67(2):192-331. doi: 10.1016/j.ejvs.2023.11.002. Epub 2024 Jan 23. PMID 38307694
- [Background] Dewulf M, Muysoms F, Vierendeels T, Huyghe M, Miserez M, Ruppert M, Tollens T, van Bergen L, Berrevoet F, Detry O. Prevention of Incisional Hernias by Prophylactic Mesh-augmented Reinforcement of Midline Laparotomies for Abdominal Aortic Aneurysm Treatment: Five-year Follow-up of a Randomized Controlled Trial. Ann Surg. 2022 Oct 1;276(4):e217-e222. doi: 10.1097/SLA.0000000000005545. Epub 2022 Jun 28. PMID 35762612
- [Background] Muysoms FE, Detry O, Vierendeels T, Huyghe M, Miserez M, Ruppert M, Tollens T, Defraigne JO, Berrevoet F. Prevention of Incisional Hernias by Prophylactic Mesh-augmented Reinforcement of Midline Laparotomies for Abdominal Aortic Aneurysm Treatment: A Randomized Controlled Trial. Ann Surg. 2016 Apr;263(4):638-45. doi: 10.1097/SLA.0000000000001369. PMID 26943336
- [Background] Bali C, Papakostas J, Georgiou G, Kouvelos G, Avgos S, Arnaoutoglou E, Papadopoulos G, Matsagkas M. A comparative study of sutured versus bovine pericardium mesh abdominal closure after open abdominal aortic aneurysm repair. Hernia. 2015 Apr;19(2):267-71. doi: 10.1007/s10029-014-1262-4. Epub 2014 May 13. PMID 24820007
- [Background] Bevis PM, Windhaber RA, Lear PA, Poskitt KR, Earnshaw JJ, Mitchell DC. Randomized clinical trial of mesh versus sutured wound closure after open abdominal aortic aneurysm surgery. Br J Surg. 2010 Oct;97(10):1497-502. doi: 10.1002/bjs.7137. PMID 20603858
- [Background] Timmermans L, Eker HH, Steyerberg EW, Jairam A, de Jong D, Pierik EG, Lases SS, van der Ham AC, Dawson I, Charbon J, Schuhmacher C, Izbicki JR, Neuhaus P, Knebel P, Fortelny R, Kleinrensink GJ, Jeekel J, Lange JF. Short-term results of a randomized controlled trial comparing primary suture with primary glued mesh augmentation to prevent incisional hernia. Ann Surg. 2015 Feb;261(2):276-81. doi: 10.1097/SLA.0000000000000798. PMID 24983993
- [Background] Jairam AP, Timmermans L, Eker HH, Pierik REGJM, van Klaveren D, Steyerberg EW, Timman R, van der Ham AC, Dawson I, Charbon JA, Schuhmacher C, Mihaljevic A, Izbicki JR, Fikatas P, Knebel P, Fortelny RH, Kleinrensink GJ, Lange JF, Jeekel HJ; PRIMA Trialist Group. Prevention of incisional hernia with prophylactic onlay and sublay mesh reinforcement versus primary suture only in midline laparotomies (PRIMA): 2-year follow-up of a multicentre, double-blind, randomised controlled trial. Lancet. 2017 Aug 5;390(10094):567-576. doi: 10.1016/S0140-6736(17)31332-6. Epub 2017 Jun 20. PMID 28641875
- [Background] Van den Dop LM, Sneiders D, Yurtkap Y, Werba A, van Klaveren D, Pierik REGJM, Reim D, Timmermans L, Fortelny RH, Mihaljevic AL, Kleinrensink GJ, Tanis PJ, Lange JF, Jeekel J; PRIMA Trialist Group. Prevention of incisional hernia with prophylactic onlay and sublay mesh reinforcement vs. primary suture only in midline laparotomies (PRIMA): long-term outcomes of a multicentre, double-blind, randomised controlled trial. Lancet Reg Health Eur. 2023 Nov 22;36:100787. doi: 10.1016/j.lanepe.2023.100787. eCollection 2024 Jan. PMID 38188275
- [Background] Hew CY, Rais T, Antoniou SA, Deerenberg EB, Antoniou GA. Prophylactic Mesh Reinforcement Versus Primary Suture for Abdominal Wall Closure after Elective Abdominal Aortic Aneurysm Repair with Midline Laparotomy Incision: Updated Systematic Review Including Time-To-Event Meta-Analysis and Trial Sequential Analysis of Randomized Controlled Trials. Ann Vasc Surg. 2024 Dec;109:149-161. doi: 10.1016/j.avsg.2024.06.026. Epub 2024 Jul 16. PMID 39025216
- [Background] Indrakusuma R, Jalalzadeh H, van der Meij JE, Balm R, Koelemay MJW. Prophylactic Mesh Reinforcement versus Sutured Closure to Prevent Incisional Hernias after Open Abdominal Aortic Aneurysm Repair via Midline Laparotomy: A Systematic Review and Meta-Analysis. Eur J Vasc Endovasc Surg. 2018 Jul;56(1):120-128. doi: 10.1016/j.ejvs.2018.03.021. Epub 2018 Apr 22. PMID 29685678
- [Background] Nicolajsen CW, Eldrup N. Abdominal Closure and the Risk of Incisional Hernia in Aneurysm Surgery - A Systematic Review and Meta-analysis. Eur J Vasc Endovasc Surg. 2020 Feb;59(2):227-236. doi: 10.1016/j.ejvs.2019.07.041. Epub 2020 Jan 3. PMID 31911135
- [Background] Tansawet A, Numthavaj P, Techapongsatorn S, Wilasrusmee C, Attia J, Thakkinstian A. Mesh position for hernia prophylaxis after midline laparotomy: A systematic review and network meta-analysis of randomized clinical trials. Int J Surg. 2020 Nov;83:144-151. doi: 10.1016/j.ijsu.2020.08.059. Epub 2020 Sep 12. PMID 32927135
- [Background] Aiolfi A, Cavalli M, Gambero F, Mini E, Lombardo F, Gordini L, Bonitta G, Bruni PG, Bona D, Campanelli G. Prophylactic mesh reinforcement for midline incisional hernia prevention: systematic review and updated meta-analysis of randomized controlled trials. Hernia. 2023 Apr;27(2):213-224. doi: 10.1007/s10029-022-02660-4. Epub 2022 Aug 3. PMID 35920944
- [Background] Tansawet A, Numthavaj P, Techapongsatorn S, McKay G, Attia J, Pattanaprateep O, Thakkinstian A. Risk-benefit assessment of onlay and retrorectus mesh augmentation for incisional hernia prophylaxis: A secondary analysis from network meta-analysis. Int J Surg. 2021 Aug;92:106053. doi: 10.1016/j.ijsu.2021.106053. Epub 2021 Aug 8. PMID 34375768
- [Background] Fischer JP, Basta MN, Wink JD, Krishnan NM, Kovach SJ. Cost-utility analysis of the use of prophylactic mesh augmentation compared with primary fascial suture repair in patients at high risk for incisional hernia. Surgery. 2015 Sep;158(3):700-11. doi: 10.1016/j.surg.2015.02.030. Epub 2015 Jul 15. PMID 26189071
- [Background] Lima HVG, Rasslan R, Novo FCF, Lima TMA, Damous SHB, Bernini CO, Montero EFS, Utiyama EM. Prevention of Fascial Dehiscence with Onlay Prophylactic Mesh in Emergency Laparotomy: A Randomized Clinical Trial. J Am Coll Surg. 2020 Jan;230(1):76-87. doi: 10.1016/j.jamcollsurg.2019.09.010. Epub 2019 Oct 28. PMID 31672681
- [Background] Jakob MO, Haltmeier T, Candinas D, Beldi G. Biologic mesh implantation is associated with serious abdominal wall complications in patients undergoing emergency abdominal surgery: A randomized-controlled clinical trial. J Trauma Acute Care Surg. 2020 Dec;89(6):1149-1155. doi: 10.1097/TA.0000000000002877. PMID 32649617
- [Background] Pizza F, D'Antonio D, Ronchi A, Lucido FS, Brusciano L, Marvaso A, Dell'Isola C, Gambardella C. Prophylactic sublay non-absorbable mesh positioning following midline laparotomy in a clean-contaminated field: randomized clinical trial (PROMETHEUS). Br J Surg. 2021 Jun 22;108(6):638-643. doi: 10.1093/bjs/znab068. PMID 33907800
- [Derived] Sguinzi R, Lagger M, Chevalley T, Gremaud B, Menth M, Buhler L, Adamina M. Prophylactic mesh reinforcement after open aortic aneurysm repair: a prospective cohort study. Front Surg. 2025 Nov 14;12:1658180. doi: 10.3389/fsurg.2025.1658180. eCollection 2025. PMID 41321852